CLINICAL TRIAL: NCT04715867
Title: A Double-blind Randomized, Controlled, Non-inferiority Trial to Evaluate the Immunogenicity and Safety of New Rabies Vaccine 'Rabix-VC' on Bangladeshi Healthy Adults
Brief Title: Non Inferiority Trial of Locally Manufactured Rabies Vaccine 'Rabix-VC' in Bangladesh
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-20117
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-12

CONDITIONS: Non Inferiority Trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group for intramuscular route (Experimental): 110 adult participant will get Ravix-VC
  Interventions: Drug: Rabix-VC
- Comparator group for intramuscular route (Active Comparator): 110 adult participant will get Rabipur
  Interventions: Drug: Rabix-VC
- Test Group for Intradermal Route (Experimental): 110 adult participant will get Ravix-VC
  Interventions: Drug: Rabix-VC
- Comparator Group for Intradermal Route (Active Comparator): 110 adult participant will get Rabipur
  Interventions: Drug: Rabix-VC

INTERVENTIONS:
Drug: Rabix-VC — Rabix-VC will be locally manufactured by Incepta Vaccine Ltd
  Other Names: Rabipur

SUMMARY:
Rabies is a viral infectious disease of mammals including humans. Early symptoms of rabies include fever and tingling at the site of exposure, followed by one or more symptoms such as fear of water, violent movements, confusion, uncontrolled excitement, inability to move parts of the body, and loss of consciousness. Once symptoms of the disease develop, rabies is invariably fatal. It is one of the oldest human diseases. It continues to be a major public health problem in developing countries. Rabies is the 10th biggest cause of death due to infectious diseases worldwide. Rabies is endemic in Bangladesh with high public health significance and ranked third highest among rabies-endemic countries for human rabies deaths. In Bangladesh, an estimated 200 000 animal bite cases with more than 2000 human rabies deaths are reported annually. Most importantly, most of the victims are children below 15 years old coming from poor rural communities.

Rabies is a vaccine-preventable viral disease and is highly effective when given pre- or post-exposure to a bite from a potentially rabid animal. Currently there is no locally manufactured Rabies vaccine available in Bangladesh. The results of this study will provide information regarding the immunogenicity and safety of the locally manufactured Rabies vaccine 'Rabix VC' as a test vaccine using 'Rabipur' as a comparator vaccine in a non inferiority study design.

DETAILED DESCRIPTION:
This will be a randomized, controlled, double-blind, parallel design, comparative, non-inferiority study on a total of 440 healthy adult participants (18-75 years of age). Participants who will be eligible for the study, will be invited to participate in the study. The study will be conducted in four groups. In One Comparator group, 110 participants will receive Rabipur through Intramuscular Route, in Test group, 110 participants will receive Rabix VC through Intramuscular Route. In another Comparator group, 110 participants will receive Rabipur through Intradermal Route and Test group, 110 participants will receive Rabix VC through Intradermal Route. Total 220 participants will receive Rabix VC (Test Group) and 220 participants will receive Rabipur (Comparator Group), 1.0 ml through Intramuscular Route and 0.2 ml through Intradermal Route, (0.1 ml each arm) respectively.

Informed consent will be obtained from the participants. Only participants who give voluntary consent will be enrolled in the study. The potential risk and the procedures to be carried out are mentioned in the consent form. Compensation will include transportation costs for the participants. Participants only can decide whether they will participate in the study. They will also be able to withdraw their name from the study at any time, without giving any explanation, and will be able to refuse collection of any or all laboratory samples for the study.

Participants may not directly benefit from participating in the study; however, results obtained from this study will be useful in understanding of potential antigenic components for designing an effective Shigella vaccine and may thus benefit the society. The whole study period for each individual will be 90 days. Specimen collection and interview will be carried out 9-10 (maximum) times including enrollment and it will take around 30 minutes per visit.

After taking consent from participants, they will be asked to do the following: Blood (10-12 ml for adults) specimens will be collected at screening (day -7 to -2), day 14 and day 30 or day 44. For Intramuscular group vaccination schedule will be on day 0, day 7, day 21 and day 0, day 3, day 7, day 28 for intradermal group. Also, there will be additional follow up on day 60 and final visit on day 90.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females of age 18 years to 75 years. 2. Individuals who had given written consent. 3. Individuals in good health and available for all the visits scheduled in the study.

Exclusion Criteria:

* 1. Pregnancy or unwillingness to practice acceptable contraception. 2. A history of Rabies vaccination. 3. Known hypersensitivity to neomycin, tetracycline, amphotericin-B or any other vaccine component.

  4. A significant acute or chronic infectious disease or use of antibiotics that may impact the subject's safety and /or immunogenicity in the Investigators opinion at the time of enrolment.

  5. Body temperature ≥38.0°C (≥ 100.4°F) within 3 days of study vaccination. 6. Individuals who received any other vaccines within 28 days prior to enrolment.

  7. Clinically Significant abnormalities in screening hematology and serum bio-chemistry, as determined by the study physician.

  8. Subjects who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.

  9. Any planned surgery during the study period. 10. Subjects who have cancer disorders excluding non-melatonin skin cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of immunogenicity by Seroconversion | One year
  The test vaccine will induce similar seroconversion rates in compare to reference vaccine. This will be done by calculating the responder rate through comparing the pre, day 14 and 30 days of initial post-vaccination Rabies Neutrializing Antibody titres among 'Rabix-VC' or 'Rabipur' vaccinated participants. The non-inferiority margin will be 10 percent. Rabies virus Neutralizing Antibody Titre ≥ 0.5 IU/ml will be logarithmically transformed prior to statistical analyses in order to better approximate normality. Student's t-test will be performed for continuous outcomes. Analysis of covariance may be used to adjust for imbalances in baseline titres. No interim analysis is planned.

SECONDARY OUTCOMES:
Safety data analysis | One Year
  1. Total number and percentage of immediate reactions (adverse events) reported within 30 minutes after vaccinations.
  2. Total number and percentage of solicited adverse events (prelisted in the participant's memory aid) occurring up to 7 days following vaccination.
  3. Total number and percentage of unsolicited AEs up to 90 days after initial vaccination.
  4. Occurrence of serious adverse events (SAEs) throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Taufiqur Rahman, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddrb, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
By publication in the journal
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After completion of the study
Access Criteria: Journal